CLINICAL TRIAL: NCT04257591
Title: Effects of Hamstrings Strengthening in Proffesional Athlets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Luis Ceballos Laita, Ph.D, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI 20- 1589
Record Dates: First submitted 2020-01-31; First posted 2020-02-06 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Exercise; Hamstring Injury
Keywords: exercise; therapeutics; prevention
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hamstring strengthening (Experimental): 8-week protocol (3 days per week) based on isometric, concentric and excentric exercisesof hamstrings
  Interventions: Other: hamstring strengthening
- Control (No Intervention): No intervention added to regular training.

INTERVENTIONS:
Other: hamstring strengthening — A progressive and individualized hamstring strengthening protocol
  Arms: hamstring strengthening

SUMMARY:
Athelts that meet the inclusion criteria will be randomized into two groups. The experimental group will receive an 8-week (3 days per week) specificl protocol based on hamstring strengthening (isometric, concentric and excentric exercises), and the control group will not receive any additional exercise. The aim of the study is to investigate the changes in hip and knee muscle strength, in the extensibility of cuadriceps, hamstrings and hip abductors, in the physical functions and in the final marks.

ELIGIBILITY:
Inclusion Criteria:

* Professional Athlet
* 3 or more trainign days
* Previous hamstring injury but without symptoms for 3 months or >30% difference between cuadriceps and hamstrings strength (considered as a risk for hamstring injury)

Exclusion Criteria:

* Sistemic pathologies
* Any other type of musculoskeletal injuries in lower limb or lumbar spine
* To have a previous specific protocol
* To skip more than 3 training days
* General contraindications for physical activity

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
muscle strength | Baseline
  the examiners assess the muscle strength using a hand-held dynamometer (model 01165) for hip and knee muscles
muscle strength | up to 8 weeks
  the examiners assess the muscle strength using a hand-held dynamometer (model 01165) for hip and knee muscles
muscle extensibility | Baseline
  the examiners assess the extensibility of the hip flexors, abductors and extensor muscles
muscle extensibility | up to 8 weeks
  the examiners assess the extensibility of the hip flexors, abductors and extensor muscles

SECONDARY OUTCOMES:
Physical function | Baseline
  the examiners assess the physical function using vertical jump test
Physical function | up to 8 weeks
  the examiners assess the physical function using vertical jump test
Mark | Baseline
  the examiners assess the marks in competition
Mark | up to 8 weeks
  the examiners assess the marks in competition
Number of hamstring injuries | Baseline
  the examiners assess the number of hamstring injuries
Number of hamstring injuries | up to 8 weeks
  the examiners assess the number of hamstring injuries

CONTACTS AND LOCATIONS:
Locations (1):
- Luis Ceballos Laita, Zaragoza, Spain